CLINICAL TRIAL: NCT00454766
Title: Evaluating Materials to Educate Patients About Cervical Dysplasia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1014
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Education; Cervical Dysplasia
Keywords: Patient Education; Cervical Dysplasia; Questionnaire
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Questionnaire Regarding Tailored Educational Materials
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Survey of two educational brochures with approximately the same information, but which vary in their health literacy (readability) level.
  Other Names: Survey

SUMMARY:
Primary Objective:

To pilot test high and low literacy patient education materials for colposcopy clinic patients, assessing impact on patient knowledge and patient feedback about the materials.

DETAILED DESCRIPTION:
Women with an abnormal Papanicolaou (Pap) smear are typically referred for a colposcopy and biopsy. However, data collected by research groups and others shows that women with abnormal Pap smear results have limited understanding of the meaning of the results, the causes of cervical dysplasia, and the procedures used to evaluate and treat it. This situation is further complicated by the fact that many patients, particularly those with less education, have low health literacy in general. This means that much of the existing patient education materials will likely be inappropriate or ineffective for this group. One approach is to develop materials at low literacy levels; however, it is not known whether such materials will be provide sufficient information and be effective for patients with high health literacy.

The long term goal is to study the importance of tailoring patient education materials to colposcopy patients' level of health literacy. To this end, researchers have developed two educational brochures with approximately the same information, but which vary in their health literacy (readability) level. As a first step in this research, researchers propose to present these materials to colposcopy patients returning for colposcopy visits to assess changes in knowledge and obtain patient feedback on the brochures.

The proposed pilot study represents the first step at evaluating the patient education materials and determining the patient's level of understanding of what they receive.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old;
2. Follow up colposcopy clinic patients who completed a colposcopy and treatment (if indicated) at an earlier date;
3. Able to communicate in English

Exclusion Criteria: None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women, over 18 years of age, with an abnormal Papanicolaou (Pap) smear are referred for a colposcopy and biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-02 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
To study the importance of tailoring patient education materials to colposcopy patients' level of health literacy. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Karen Basen-Engquist, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org